CLINICAL TRIAL: NCT07013071
Title: The Effect of Different Vasoconstrictive Agents on Hemodynamics Among Patients Undergoing Simple Mandibular Exodontia: A Triple-Blind Randomized Controlled Trial
Brief Title: Hemodynamic Effects of Different Vasoconstrictors in Mandibular Exodontia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Razan Baabdullah, Assistant professor of oral and maxillofacial surgery, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 240-11-23
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Hemodynamics; Pain; ASA I-II Requiring Simple Dental Extraction of a Mandibular Tooth
Keywords: Mepivacaine 2% with vasoconstrictor; Hemodynamic effects of vasoconstrictors; Epinephrine vs epinephrine bitartrate; Pain control during dental extraction; Blood pressure and heart rate during dental procedures
MeSH Terms: conditions — Pain | interventions — Mepivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: This study used a triple-blind, parallel assignment randomized controlled trial design. Participants were randomly assigned to one of two groups: one group received 2% mepivacaine with 1:100,000 epinephrine, and the other received 2% mepivacaine with 1:55,000 epinephrine bitartrate. Both groups underwent simple mandibular tooth extraction, and their hemodynamic responses and pain levels were assessed at standardized intervals. The study maintained blinding across patients, care providers, and outcome assessors to minimize bias.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epinephrine Group (1:100,000) (Active Comparator): Participants in this group received local anesthesia consisting of 2% mepivacaine hydrochloride with 1:100,000 (0.01 mg/mL) epinephrine prior to simple mandibular tooth extraction. This arm served as the comparator for evaluating hemodynamic changes and pain control.
  Interventions: Drug: 2% Mepivacaine with 1:100,000 epinephrine
- Epinephrine Bitartrate Group (1:55,000) (Experimental): Participants in this group received local anesthesia consisting of 2% mepivacaine hydrochloride with 1:55,000 (0.018 mg/mL) epinephrine bitartrate prior to simple mandibular tooth extraction. This arm was evaluated for its effects on hemodynamic parameters and pain perception compared to standard epinephrine.
  Interventions: Drug: 2% Mepivacaine with 1:55,000 Epinephrine Bitartrate

INTERVENTIONS:
Drug: 2% Mepivacaine with 1:100,000 epinephrine — A standard vasoconstrictor-containing local anesthetic used in dental procedures to minimize bleeding and prolong anesthetic effect.
  Arms: Epinephrine Group (1:100,000)
Drug: 2% Mepivacaine with 1:55,000 Epinephrine Bitartrate — An alternative formulation of vasoconstrictor-containing local anesthetic evaluated for its safety and analgesic effectiveness in dental extractions.
  Arms: Epinephrine Bitartrate Group (1:55,000)

SUMMARY:
Title of Study:

The Effect of Different Vasoconstrictive Agents on Hemodynamics Among Patients Undergoing Simple Mandibular Exodontia: A Triple-Blind Randomized Controlled Trial

Location:

King Abdulaziz University Dental Hospital (KAUFD), Jeddah, Saudi Arabia What Is This Study About?

This study examines two types of vasoconstrictive agents used alongside local anesthetic during simple lower tooth extractions:

* Epinephrine (1:100,000)
* Epinephrine Bitartrate (1:55,000)

What are vasoconstrictors? Vasoconstrictors help control bleeding and extend the numbing effect during dental procedures. They are usually added to local anesthetics (numbing agent) during dental procedures. This research aims to answer the following questions:

1. Which one of the vasoconstrictive agents has less effect on the heart rate and blood pressure
2. Which one offers better pain control?

Who Can participate?

* Adult patient +18 year/old or above (healthy or with well-controlled conditions like hypertension)
* Patients who require non-surgical lower tooth extractions
* Procedures will be done by supervised fifth and sixth-year dental students

Potential Risks and Discomforts

Like any medical procedure, there are some potential risks, including:

From the anesthesia and vasoconstrictors:

* Allergic reaction
* Prolonged numbness
* Changes in blood pressure and heart rate

From the tooth extraction itself:

* Bleeding
* Pain or discomfort
* Swelling or bruising
* Infection
* Dry socket
* Delayed healing
* Damage to nearby teeth or tissues
* Fracture of the tooth or jawbone
* Numbness or altered sensation (temporary or permanent)
* Sinus complications (in upper tooth extractions)
* The need for additional procedures

Potential Benefits

* Free tooth extraction
* Blood pressure monitoring - with referral to a primary care provider if undiagnosed high blood pressure is detected

Costs There are no additional costs to participate in this research. Treatment and extraction are provided free of charge.

Compensation / Treatment for Injury

If a participant is injured as a result of being in this study:

* Necessary treatment and medical care will be provided by the research team.
* No financial compensation is available from King Abdulaziz University Dental Hospital (KAUFD).

Confidentiality Participants' identity and medical information will be kept confidential. Only authorized researchers and relevant oversight bodies may access Participants' medical/dental records for monitoring or auditing purposes, in accordance with laws and regulations. Any published results will not identify the participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* ASA I or II classification (i.e., healthy or with mild systemic disease).
* Requiring simple mandibular tooth extraction, as defined by painless removal with minimal tissue trauma and smooth postoperative healing.
* Willing and able to provide informed consent.
* Able to comply with study procedures (able to undergo the simple tooth extraction).

Exclusion Criteria:

* Pregnant or lactating individuals.
* ASA III or higher classification (i.e., patients with severe systemic disease).
* Patients with uncontrolled systemic disease.
* History of malignancy.
* Presence of unstable psychiatric illness.
* Current use of antiplatelet or anticoagulant medications.
* Known allergies to local anesthetics.
* Uncooperative patients or those with intellectual disabilities.
* Cases requiring surgical extractions (e.g., needing tooth sectioning, mucoperiosteal flaps, or bone removal).
* Patients requiring maxillary tooth extraction.
* Presence of fascial space infection or acute oral conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Change in Systolic and Diastolic Blood Pressure | Measured preoperatively, 3 minutes post-anesthesia (intraoperative), and immediately after the procedure (postoperative).
  To compare changes in systolic and diastolic blood pressure between the two groups (epinephrine vs. epinephrine bitartrate) at three time points: before administration of local anesthesia, 3 minutes after administration (intraoperative), and postoperatively following simple mandibular tooth extraction.
Change in Heart Rate | Measured preoperatively, 3 minutes post-anesthesia (intraoperative), and immediately after the procedure (postoperative).
  To evaluate changes in heart rate between the two intervention groups across the same three time points to assess the hemodynamic impact of the vasoconstrictors used.

SECONDARY OUTCOMES:
Pain Score Using Visual Analogue Scale (VAS) | Assessed every 30 minutes during the procedure and once at the completion of the extraction.
  To compare pain perception during and after the dental procedure between the two groups using a 10-point Visual Analogue Scale (VAS). Patients reported pain at 30-minute intervals throughout the procedure and at the end of treatment. The minimum value on the VAS is 0 and the maximum is 10.

CONTACTS AND LOCATIONS:
Overall Officials: Razan M Baabdullah, BDS, MS, FRCDC, Principal Investigator — King Abdulaziz University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery
Locations (1):
- King Abdulaziz University, Faculty of Dentistry, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Karm MH, Park FD, Kang M, Kim HJ, Kang JW, Kim S, Kim YD, Kim CH, Seo KS, Kwon KH, Kim CH, Lee JW, Hong SW, Lim MH, Nam SK, Cho JM. Comparison of the efficacy and safety of 2% lidocaine HCl with different epinephrine concentration for local anesthesia in participants undergoing surgical extraction of impacted mandibular third molars: A multicenter, randomized, double-blind, crossover, phase IV trial. Medicine (Baltimore). 2017 May;96(21):e6753. doi: 10.1097/MD.0000000000006753. PMID 28538371
- [Result] Gupte SH, Kalra RD, Dcruz TM, Kamble S, Patnaik RS. Comparative Evaluation of Effectiveness of 2% Lignocaine Hydrochloride with Clonidine Hydrochloride versus 2% Lignocaine Hydrochloride with Adrenaline Bitartrate as Local Anesthetic for Adult Patients Undergoing Surgical Extraction of Impacted Mandibular Third Molars: A Randomized Controlled Clinical Study. Contemp Clin Dent. 2021 Jul-Sep;12(3):308-312. doi: 10.4103/ccd.ccd_665_20. Epub 2021 Sep 21. PMID 34759690
- [Result] Abu-Mostafa N, Al-Showaikhat F, Al-Shubbar F, Al-Zawad K, Al-Zawad F. Hemodynamic changes following injection of local anesthetics with different concentrations of epinephrine during simple tooth extraction: A prospective randomized clinical trial. J Clin Exp Dent. 2015 Oct 1;7(4):e471-6. doi: 10.4317/jced.52321. eCollection 2015 Oct. PMID 26535092
- [Result] Conrado VC, de Andrade J, de Angelis GA, de Andrade AC, Timerman L, Andrade MM, Moreira DR, Sousa AG, Sousa JE, Piegas LS. Cardiovascular effects of local anesthesia with vasoconstrictor during dental extraction in coronary patients. Arq Bras Cardiol. 2007 May;88(5):507-13. doi: 10.1590/s0066-782x2007000500002. English, Portuguese. PMID 17589623
- [Result] Silvestre FJ, Martinez-Herrera M, Garcia-Lopez B, Silvestre-Rangil J. Influence of anxiety and anesthetic vasoconstrictors upon hemodynamic parameters during dental procedures in controlled hypertensive and non-hypertensive patients. J Clin Exp Dent. 2021 Feb 1;13(2):e156-e164. doi: 10.4317/jced.57232. eCollection 2021 Feb. PMID 33575000
- [Result] Seminario-Amez M, Gonzalez-Navarro B, Ayuso-Montero R, Jane-Salas E, Lopez-Lopez J. USE OF LOCAL ANESTHETICS WITH A VASOCONSTRICTOR AGENT DURING DENTAL TREATMENT IN HYPERTENSIVE AND CORONARY DISEASE PATIENTS. A SYSTEMATIC REVIEW. J Evid Based Dent Pract. 2021 Jun;21(2):101569. doi: 10.1016/j.jebdp.2021.101569. Epub 2021 Apr 10. PMID 34391560
- [Result] Ezmek B, Arslan A, Delilbasi C, Sencift K. Comparison of hemodynamic effects of lidocaine, prilocaine and mepivacaine solutions without vasoconstrictor in hypertensive patients. J Appl Oral Sci. 2010 Jul-Aug;18(4):354-9. doi: 10.1590/s1678-77572010000400006. PMID 20835569
- [Result] Tsuchihashi T, Takata Y, Kurokawa H, Miura K, Maruoka Y, Kajiyama M, Fujishima M. Blood pressure response during dental surgery. Hypertens Res. 1996 Sep;19(3):189-94. doi: 10.1291/hypres.19.189. PMID 8891747
- [Result] Silvestre FJ, Salvador-Martinez I, Bautista D, Silvestre-Rangil J. Clinical study of hemodynamic changes during extraction in controlled hypertensive patients. Med Oral Patol Oral Cir Bucal. 2011 May 1;16(3):e354-8. doi: 10.4317/medoral.16.e354. PMID 21196862
- [Result] Abhijith George, Mandeep Sharma, Prasanna Kumar, Sneha Kulkarni, Vinay Patil y Jacob John Plackal. Hemodynamic changes during exodontia in hypertensive and normotensive patients following injection of local anesthetics with and without epinephrine: a prospective comparative study. Rev Esp Cir Oral Maxilofac. 2022;44(1):9-15.
- [Result] Ogunlewe MO, James O, Ajuluchukwu JN, Ladeinde AL, Adeyemo WL, Gbotolorun OM. Evaluation of haemodynamic changes in hypertensive patients during tooth extraction under local anaesthesia. West Indian Med J. 2011 Jan;60(1):91-5. PMID 21809720
- [Result] Matsumura K, Miura K, Takata Y, Kurokawa H, Kajiyama M, Abe I, Fujishima M. Changes in blood pressure and heart rate variability during dental surgery. Am J Hypertens. 1998 Nov;11(11 Pt 1):1376-80. doi: 10.1016/s0895-7061(98)00157-5. PMID 9832183

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT07013071/Prot_SAP_000.pdf